CLINICAL TRIAL: NCT02737852
Title: A Single-Center, Clinical Study to Evaluate the Safety of a New Personal Lubricant in Healthy Female Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ST-7609
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Erythema; Edema
MeSH Terms: conditions — Erythema; Edema

STUDY DESIGN:
Masking Description: The new personal lubricant was used by all participants

ARMS (1):
- Healthy subject (Experimental): Healthy subject exposed to Trojan "Chameleon" Personal Lubricant at least four times weekly for two weeks
  Interventions: Device: Trojan "Chameleon" Personal Lubricant

INTERVENTIONS:
Device: Trojan "Chameleon" Personal Lubricant — silicone base with sensate

SUMMARY:
To evaluate the safety of a new personal lubricant when used at least four times weekly for two weeks (including at least twice weekly during sexual intercourse for subjects with monogamous male partners), in a population consisting of healthy females.

ELIGIBILITY:
Inclusion Criteria:

* no participation in a similar study 2-weeks prior
* may be post-menopausal or have had a hysterectomy
* if sexually active, and of child bearing potential, subjects using adequate non-barrier method of birth control
* free from any vaginal disorders
* sexually active and monogamous, heterosexual relationship, and whose male partner is willing and able to give informed consent and agrees to engage in sexual intercourse at least twice each week during the two-week study or is not sexually active
* personal lubricant user and agrees to replace her usual personal lubricant with the investigational product
* can start regardless of where they are in their cycles
* agrees to use the provided investigational product at least four times weekly over the two week study period
* exhibits no clinically significant evidence of vulvar or vaginal irritation, as determined by a study doctor, and no reports of sensory irritation at the baseline exam
* willing to refrain from introducing any new vaginal products, or using vaginal medications or local contraceptives during study
* agrees to refrain from douching or using any medications, powder, lotions or personal care products in the vulvar or perianal area
* willing to use a urine pregnancy test provided to them at baseline and on third visit
* standard medical history form on file
* signed informed consent
* completed HIPAA
* dependable and able to follow directions as outlined
* receives a score of 0 or 0.5 for erythema and edema: and 0 for sensorial irritation (burning, stinging, itching and dryness) during the first examination.

Exclusion Criteria:

* pregnant, nursing or planning a pregnancy
* currently using or has used within two weeks prior to the study initiation, any systemic or topical corticosteroids, vasoconstrictors, antibiotics, anti-inflammatories or antihistamines
* known allergies to vaginal or any cosmetic products
* reports history of recurrent bladder, vaginal infections or incontinence
* exhibits or reports gynecologic abnormalities or has had vaginitis within 60 days prior to study initiation
* uses a vaginal ring, diaphram or cervical/vault caps, condoms, or condoms with spermicide as a means of contraception
* participated in a study involving the vaginal area or in an investigational systemic drug study within two weeks of study initiation
* receives a score higher than 0/5 for erythema, edema or >0 for burning, stinging, or itching, during first examination or shows any other sign of mucosal irregularities

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Laboratories, LLC, Piscataway, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Subject
Started | 32
Completed | 30
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Subject
Number analyzed (Participants) | 30
Age, Customized [Count of Participants; unit: Participants]
  Age 19-59 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Observed Local Erythema Based on the 5 Point Scoring Scale
Description: Number of subjects with observed local erythema by obstetrician/gynecologist examination as graded on 5 point clinical scale: 0 = normal appearance no irritation, 0.5 = slight, irregular erythema, 1 = mild erythema, 2 = moderate erythema 3 = severe erythema
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Subject
Number analyzed (Participants) | 30
Participants | 0

2. Primary Outcome: Number of Subjects With Observed Edema Based on the 5 Point Scoring Scale
Description: Number of subjects with observed local edema by obstetrician/gynecologist examination as graded on 5 point clinical scale: 0 = normal appearance no edema, 0.5 = slight edema, 1 = mild edema, 2 = moderate edema 3 = severe edema
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Subject
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Arm/Group | Healthy Subject
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Master service agreement and confidentiality agreement in place